CLINICAL TRIAL: NCT01473602
Title: Second Study of the Effect of Teriparatide on Femoral Neck Fracture Healing
Brief Title: Second Study of the Effect of Teriparatide on Hip Fracture Healing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14125; B3D-MC-GHDQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Femur Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Administered once daily by subcutaneous (SC) injection for 6 months
  Interventions: Drug: Placebo; Dietary Supplement: Calcium supplementation; Dietary Supplement: Vitamin D supplementation
- Teriparatide (Experimental): 20 microgram (µg) administered once daily by SC injection for 6 months
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium supplementation; Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Drug: Teriparatide — Administered by SC injection
  Other Names: Forteo; Forsteo; LY333334
  Arms: Teriparatide
Drug: Placebo — Administered by SC injection
  Arms: Placebo
Dietary Supplement: Calcium supplementation — Administered orally
Dietary Supplement: Vitamin D supplementation — Administered orally

SUMMARY:
The purpose of this study is to see whether teriparatide, given for 6 months versus placebo, will improve the healing of hip (femoral neck) fractures that are repaired during surgery using certain types of orthopedic screws. The study will enroll men and postmenopausal women at least 50 years of age with a recent hip (femoral neck) fracture caused by low-trauma (for example, fall from standing height or less).

DETAILED DESCRIPTION:
This is a 12-month, Phase 3, prospective, randomized, parallel, double-blind, placebo-controlled, multicenter, multinational study to evaluate the effect of 6 months of treatment with teriparatide on fracture healing in participants who have sustained a recent low-trauma, unilateral, femoral neck fracture stabilized by internal fixation. The study has 3 periods:

1. A screening period that must be completed in ≤ 14 days after operative treatment of the femoral neck fracture
2. A 6-month double-blind treatment period [teriparatide 20 (µg) or placebo given once daily by subcutaneous injection]
3. A 6-month observation period.

The primary objective is to assess the effect of 6 months of treatment with teriparatide 20 µg/day versus placebo on the proportion of men and postmenopausal women of at least 50 years of age with no revision surgery 12 months after internal fixation of a low-trauma femoral neck fracture.

All participants will receive supplements of calcium and vitamin D beginning at screening and continuing for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and postmenopausal women who were ambulatory before sustaining a low-trauma, unilateral femoral neck fracture (displaced or nondisplaced)
* Other than femoral neck fracture, be free of incapacitating conditions and have a life expectancy of at least 2 years
* Have received or are eligible for treatment with internal fixation (sliding hip screw or multiple cancellous screws) for the femoral neck fracture (the surgical procedure itself is not performed as part of this study)
* Have given written informed consent (participant or proxy) after being informed of the risks, medications, and study procedures

Exclusion Criteria:

* Increased baseline risk of osteosarcoma
* History of unresolved skeletal diseases affecting bone metabolism other than primary osteoporosis
* Abnormally elevated serum calcium at screening
* Abnormally elevated serum intact parathyroid hormone (PTH) (1-84) at screening
* Severe vitamin D deficiency at screening
* Active liver disease or jaundice
* Significantly impaired renal function
* Abnormal thyroid function not corrected by therapy
* History of malignant neoplasm in the 5 years prior to screening
* History of bone marrow or solid organ transplantation
* History of symptomatic nephrolithiasis or urolithiasis in the 1 year prior to screening
* Previous treatment with the following bone active drugs is allowed but must be discontinued at screening: oral bisphosphonates, selective estrogen receptor modulators (SERMs), calcitonin, estrogen (oral, transdermal, or injectable), progestin, estrogen analog, estrogen agonist, estrogen antagonist or tibolone, and active vitamin D3 analogs. Androgen or other anabolic steroid use must be discontinued, except for use of physiologic replacement testosterone
* Previous treatment with the following bone active drugs is exclusionary, if the stated treatment durations have been met: strontium ranelate for any duration, intravenous bisphosphonates in the 12 months preceding screening, and/or denosumab in the 6 months preceding screening
* Prior treatment with PTH, teriparatide, or other PTH analogs, or prior participation in any other clinical trial studying PTH, teriparatide, or other PTH analogs
* Local or systemic treatment with bone morphogenic proteins or any other growth factor
* Previous fracture(s) or bone surgery in the currently fractured hip
* Soft-tissue infection at the operation site
* Treatment with bone grafting or osteotomies
* Treatment with augmentation using any type of degradable cement, hydroxyapatite-coated implants, or with noninvasive interventions
* Associated major injuries of a lower extremity including fractures of the foot, ankle, tibia, fibula, knee, femur, femoral head, or pelvis; dislocations of the ankle, knee, or hip

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Golden, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockford, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falls Church, Virginia
- Belgium (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Blankenberge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Croatia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sisak
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari/Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eger
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hatvan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
- India (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Attavar, Mangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Switzerland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lausanne
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Teriparatide 20 microgram (µg) once-daily by subcutaneous (SC) injection for 6 months. Participants received calcium and vitamin D supplements.
- Placebo: Placebo once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
Period: Overall Study
Arm/Group | Teriparatide | Placebo
Started | 18 | 21
Received at Least 1 Dose of Study Drug | 18 | 20
Completed 6 Months | 12 | 15
Completed 12 Months | 10 | 13
Completed | 10 | 13
Not Completed | 8 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Groups:
- Teriparatide: Teriparatide 20 µg once-daily by subcutaneous (SC) injection for 6 months. Participants received calcium and vitamin D supplements.
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Placebo | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.39 (10.259) | 69.93 (10.417) | 71.57 (10.351)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
  Hungary | 6 | 8 | 14
  Belgium | 2 | 1 | 3
  Romania | 2 | 3 | 5
  Netherlands | 2 | 2 | 4
  Korea, Republic of | 4 | 5 | 9
Surgical screw type [Number; unit: participants] — Surgical screws used in initial surgery to repair femur neck hip fracture.
  participants
    Cancellous Screws | 18 | 18 | 36
    Sliding Hip Screws | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Revision Surgery at 12 Months After Internal Fixation of a Low-Trauma Femoral Neck Fracture
Description: Revision surgery (re-operation) was defined as any additional surgical intervention performed or recommended at the site of the index procedure, except those that were planned at the time of the index procedure.
Time Frame: 12 months
Population: Participants who were randomized, received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Percentage of participants | 74 [51 to 88] | 93 [70 to 99]

2. Secondary Outcome: Percentage of Participants With Radiographic Evidence of Healing
Description: The signs of femoral neck fracture healing and healing complications included disappearance of the fracture line on radiographs. If a participant had radiographic evidence of healing at the 12-month visit, that participant was considered to have radiographic evidence of healing.
  Percentage was calculated as: (number of participants with radiographic evidence of healing / total number of participants analyzed) * 100.
Time Frame: Randomization up to 12 months
Population: Participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Percentage of participants | 55.6 | 65.0

3. Secondary Outcome: Percentage of Participants With Pain Control During Ambulation
Description: The worst pain numeric rating scale (NRS) was used to assess the impact of pain on a participant's life. NRS Item 3 assessed the worst musculoskeletal pain severity during the walking test. Pain was measured by an 11-point Likert scale. The following cut-points were used to categorize the NRS responses: 0 = no pain, 1 to 4 = mild pain, 5 to 6 = moderate pain, and 7 to 10 = severe pain. Higher scores indicated more severe pain. Participants with an NRS score of <7 and no worsening of NRS scores >2 from baseline were categorized as having no severe fracture-site pain. Percentage was calculated as: (number of participants with pain control during ambulation / total number of participants analyzed) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug, had baseline and at least 1 nonmissing post-baseline measurement. Last observation carried forward (LOCF) values used.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 10 | 13
Percentage of participants | 90.0 | 100.0

4. Secondary Outcome: Percentage of Participants Without Severe Fracture-Site Pain During 24 Hours Prior to Visit
Description: The NRS was used to assess the impact of pain on a participant's life. Fracture-site pain severity was assessed for pain in the 24 hours preceding a visit. Pain was measured by an 11-point Likert scale. Participants with an NRS score of <7 in the 24 hours preceding a visit and no worsening of NRS score >2 from baseline were categorized as having no severe fracture-site pain. Percentage was calculated as: (number of participants with pain control during 24 hours preceding a visit / total number of participants analyzed) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug and had baseline and at least one nonmissing post-baseline measurement for severe fracture-site pain in the last 24 hours.. LOCF values used.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 11 | 14
Percentage of participants | 81.8 | 92.9

5. Secondary Outcome: Percentage of Participants Without Severe Fracture-Site Pain During Weight Bearing
Description: The worst pain NRS was used to assess the impact of pain on a participant's life. Fracture-site pain severity was assessed for pain on weight bearing. Pain was measured by an 11-point Likert scale. Participants with an NRS score of <7 during weight bearing and no worsening of NRS score >2 from baseline were categorized as having no severe fracture-site pain. Percentage was calculated as: (number of participants with pain control during weight bearing / total number of participants) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug and had baseline and at least one nonmissing post-baseline measurement. LOCF values used.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 11 | 13
Percentage of participants | 90.9 | 84.6

6. Secondary Outcome: Percentage of Participants With Functional Evidence of Healing
Description: Functional healing was defined as ability to walk with a gait speed ≥ 0.05 meters/second (m/s) with a change from baseline ≥ -0.1 m/s. The walking test involved having the participant walk a distance of 7 meters (m) at a self-selected, comfortable pace. A 4-m portion of the test was timed to determine the participant's gait speed in m/s.
  Percentage was calculated as: (number of participants with functional evidence of healing / total number of participants analyzed) * 100.
Time Frame: Up to 12 Months
Population: Participants who were randomized, received at least 1 dose of study drug, and had either at least one nonmissing gait speed or non-ambulatory status. LOCF values used.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 13 | 15
Percentage of participants | 76.9 | 66.7

7. Secondary Outcome: Percentage of Participants Able to Ambulate
Description: Ability to ambulate was defined as ambulatory with or without convalescent aid. Percentage was calculated as: (number of participants able to ambulate / total number of participants analyzed) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received treatment and had at least 1 nonmissing post-baseline measurement. LOCF values used
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 13 | 15
Percentage of participants | 76.9 | 93.3

8. Secondary Outcome: Percentage of Participants Who Regained Their Prefracture Ambulatory Status
Description: Prefracture ambulatory status was defined as either ambulatory with or without a walking aid. A participant was considered to have regained their prefracture ambulatory status if the participant's postsurgery ambulatory status was returned to or was improved from their pre-surgery ambulatory status. Percentage was calculated as = (number of participants who regained their ambulatory status / total number of participants analyzed) *100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug, and had baseline and at least one nonmissing post-baseline measurement. LOCF values used.
Measure: Number; unit: Percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 17 | 16
Percentage of participants | 47.1 | 62.5

9. Secondary Outcome: Mean Change From Baseline to 6 Months in Worst Fracture-Site Pain
Description: The worst pain NRS was used to assess the impact of pain on a participant's life. Participants with an NRS score of <7 were categorized as having no severe fracture-site pain. Least squares (LS) means was calculated using analysis of covariance (ANCOVA) adjusted for baseline, treatment group, region, fracture type, and fixation type.
Time Frame: Baseline, 6 Months
Population: Participants who were randomized, received at least 1 dose of study drug, had baseline and at least 1 nonmissing post-baseline measurement..
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale
  During ambulation ( n= 10, 13) | -1.6 (1.46) | -1.3 (1.45)
  During 24 hours preceding visit (n= 10, 14) | -1.2 (1.27) | -1.4 (1.21)
  On weight bearing (n= 10, 13) | -2.0 (1.50) | -1.4 (1.45)

10. Secondary Outcome: Mean Change From Baseline to 6 Months in Gait Speed
Description: The walking test involved having the participant walk a distance of 7 m at a self-selected, comfortable pace. A 4-m portion of the test was timed to determine the participant's gait speed in m/s. LS means was calculated using ANCOVA adjusted for baseline, treatment group, region, fracture type, and fixation type
Time Frame: Baseline, 6 Months
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 10 | 13
m/s | 0.168 (0.153) | 0.118 (0.145)

11. Secondary Outcome: Time to Revision Surgery
Description: Time to revision surgery was defined as the time from initial hip fracture surgery to revision surgery, or recommendation for revision surgery if recommended but not performed. Time to revision surgery was censored at the date of the last contact.
Time Frame: Baseline to Revision Surgery (up to 14.14 Months)
Population: Participants who were randomized, received at least 1 dose of study drug, and who did not have revision surgery or if they had revision surgery, it was adjudicated as not being related to the initial hip fracture surgery. Participants censored: Teriparatide = 14; placebo = 19.
Measure: Median (Full Range); unit: Days
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Days | 333.5 [35 to 443] | 361 [29 to 426]

12. Secondary Outcome: Mean Change From Baseline to 6 Months on Short Form-12 (SF-12) Physical (PCS) and Mental Component Summary (MCS) Scores
Description: SF-12 is a self-reported questionnaire covering a mental component score (MCS) and a physical component score (PCS), each scoring from a 0 to 100 (worst to best) scale. LS means was calculated using ANCOVA adjusted for baseline, treatment group, region, fracture type, fixation type, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 6 Months
Population: Participants who were randomized, received treatment, were adjudicated as having the hip fracture in the neck of the femur and had baseline and at least 1 nonmissing post-baseline measurement..
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale
  PCS Month 6 (n=12, 14) | 0.89 (3.0) | 1.78 (2.75)
  MCS Month 6 (n=12, 14) | -8.84 (5.80) | -10.71 (5.14)

13. Secondary Outcome: Mean Change From Baseline to 6 Months on Western Ontario McMaster Osteoarthritis Index (WOMAC)
Description: WOMAC: was a self-reported questionnaire that consisted of 24 questions covering 3 health domains: Pain (5 items: during walking, using stairs, in bed, sitting or lying, and standing), Stiffness (2 items: after first waking and later in the day), and Physical Function. Each domain was scored by summing the individual items and transforming the scores into a 0 to 100 (best to worst) scale. Lower scores indicated better health status or functioning. LS means was calculated using ANCOVA adjusted for baseline, treatment group, region, fracture type, fixation type, visit, and visit-by-treatment interaction.
Time Frame: Baseline, up to 6 Months
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale
  Physical Function Score - Month 6 (n=11, 12) | 10.5 (12.41) | 1.1 (12.42)
  Pain Score - Month 6 (n=12, 13) | 10.6 (10.64) | 13.6 (10.09)
  Stiffness Score - Month 6 (n=12, 15) | 13.5 (8.71) | 16.9 (7.74)

14. Secondary Outcome: Mean Change From Baseline to 6 Months on European Quality of Life Questionnaire (EQ-5D) Overall Health Score
Description: The EQ-5D is a 5-item, self-reported, generic, multidimensional, health-related, quality-of-life instrument with 5 items. Overall health state score was also self-reported using a visual analogue scale (VAS) marked on a scale scored from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores represented better health state with 0 representing worst imaginable health state and 100 representing best imaginable health state. LS means was calculated using ANCOVA adjusted for baseline, treatment group, region.
Time Frame: Baseline, 6 Months
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale | 13.0 (6.42) | 10.4 (6.67)

ADVERSE EVENTS:
Time Frame: Randomization to Study Completion
Groups:
- Placebo Follow-up: Follow-up after placebo once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
- Teriparatide Follow-up: Follow-up after teriparatide 20 µg once-daily by subcutaneous (SC) injection for 6 months. Participants received calcium and vitamin D supplements.
Arm/Group | Placebo | Teriparatide | Placebo Follow-up | Teriparatide Follow-up
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/18 | 3/15 | 1/12
Other Adverse Events (participants affected / at risk) | 5/20 | 3/18 | 4/15 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Teriparatide (N=18) | Placebo Follow-up (N=15) | Teriparatide Follow-up (N=12)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=20) | Teriparatide (N=18) | Placebo Follow-up (N=15) | Teriparatide Follow-up (N=12)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/16 (1) | 0/14 (0) | 0/12 (0) | 0/9 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Removal of internal fixation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days